CLINICAL TRIAL: NCT02140983
Title: Effects of Liraglutide on Hippocampal Structure and Function in Aging Adults With Prediabetes
Acronym: LGT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Natalie Rasgon, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 25076
Record Dates: First submitted 2014-01-27; First posted 2014-05-16 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Insulin Resistance; Dementia
Keywords: Insulin Resistance; Family History of Dementia; Cognition
MeSH Terms: conditions — Insulin Resistance; Dementia | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Active Comparator): 90 days of liraglutide treatment at adjusting dose, up to 1.8mg/day
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): 90 days of placebo pen, up to 1.8mg/day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — 90 days of liraglutide up to 1.8mg/day.
  Other Names: Victoza
  Arms: Liraglutide
Drug: Placebo — Placebo medication
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of liraglutide on the memory and attention of people with insulin resistance. Liraglutide is a medication that makes the body more sensitive to insulin, and therefore may allow it to manage sugar more effectively.

The investigators are looking specifically at a region of the brain that is associated with memory and attention, called the hippocampus, in order to see whether treatment this treatment will change performance on memory and attention tasks. The investigators are also taking an MRI of the brain to see whether there are changes to the size and shape of the hippocampus after treatment.

All subjects in this study will be 50-70 years old and have pre- diabetes. Half of all subjects will have a family history of dementia, while the other half will not.

DETAILED DESCRIPTION:
Data from this study will be used to measure changes in hippocampal morphology, functional alterations in the hippocampus during a paired associative memory task, functional connectivity during rest, and neuropsychological performance on hippocampally-mediated cognitive tasks, following double-blind treatment with liraglutide and placebo.

Primary Hypothesis: Subjects receive liraglutide will show significant differences in hippocampal morphology, functional activation and connectivity, and neuropsychological performance, compared to subjects receiving placebo.

Exploratory Aim: To test for potential interactions between modifiable (IR/prediabetes) and non-modifiable (FamHxAD, APOE 4) risk factors with respect to morphological, functional, and neuropshchological changes during double-blind liraglutide treatment.

Study Procedures

The study will be explained to the participant and informed consent obtained. Participant will also be asked whether or not they consent to being videotaped during the study, and if they do, parts of their study participation may be videotaped for staff training purposes. Participants will continue any current psychiatric medication(s) or psychotherapy during the duration of the study (eg. no changes will be made to currently received treatments). Psychiatric Assessment - This will consist of the Mini International Neuropsychiatric Interview(MINI), the 17-item Hamilton Depression Rating Scale (HDRS-17), and the Mini Mental Status Examination (MMSE). The MINI interview takes approximately 20-30 minutes depending on the individual presentation and has screening and skip-out questions that allow for rapid assessment of psychiatric history, current or in remission, to ensure screen-out for psychiatric exclusions.

The HDRS-17 will be used to screen out current depression, as characterized by a score of > 8. Administration of the HDRS will be repeated during and at the end of double-blind treatment. The MMSE, a brief measure of cognitive functioning that assesses arithmetic, memory and orientation, will screen out current cognitive impairment.

Physical Examination and Monitoring:

A general physical examination will be conducted at baseline and at the end of treatment. Vital signs (e.g. blood pressure, pulse, temperature, body weight) will be assessed at each in-person study visit. Individual energy (in kilocalories) expenditure per day will be assessed using self-report questionnaires (Stanford 7-Day Physical Activity Recall Scale and the Food Frequency Questionnaire).

In addition, subjects will complete the Pittsburgh Sleep Quality Index, the Memory Function Questionnaire (to assess subjective cognitive complaints) baseline and final visit, as well as report on the frequency of any alcohol or nicotine use.

All of this information will be used to adjust for differences in the experimental variables between the two experimental groups both at baseline and over the course of double-blind treatment.

Oral Glucose Tolerance Test (OGTT): After an overnight fast, subjects will be given a oral glucose challenge, wherein plasma glucose concentrations will be measured at baseline, T30min, T60min, T90min, and T120min after 75gm oral glucose load. Individuals with fasting glucose of 100-125 mg/dl and/or a 2-hour glucose of 140-199 mg/dL and less than 200 mg/dL will be eligible for study enrollment. OGTT will be repeated at the end of the study.

Oral Cortisol Swabs: The participants will be asked to take oral cortisol measures for 3 days at waking, 30 minutes after waking and at 9pm. These measures will be taken at baseline and final follow up.

Genotyping for APOE:

If the subject consents to the collection of a buffy coat sample, this will be done during the collection of blood for the blood screening tests. The amount of blood required for the buffy coat sample is approximately 2-3 teaspoons. The subject will have the right to withdraw consent for this test now or at any time and this will not affect his or her ability to participate in the research study. The sample will be stored in a minus 80 freezer for as long as, but not limited to 5 years. We will not use this sample for any other purpose without the subject's specific permission.

Genetic analysis will be conducted by experienced laboratory technicians under the supervision of Dr. Joachim Hallmayer. Blood for genotyping (approximately 6ccs) will be drawn at the time of eligibility screening, after informed consent. Genotype results will not be released to participants. Blood samples will be labeled with a unique subject identifier known only to the PI's research staff. Genotyping for APOE will be the primary genetic analysis and will be performed according to the restriction isotyping protocol of Hixson and Vernier. Two observers blind to clinical status of the individuals will carry out assignment of genotypes.

Structural and Functional MRI: Scans will be acquired on a 3.0T GE magnet at baseline and upon 12-week follow-up at the Stanford Center for Cognitive and Neurobiological Imaging (CNI). Both structural and functional brain imaging will be conducted, and total scan time will be 1 hour. All scans will be examined by a neuroradiologist to detect the presence of unanticipated structural lesions, including tumors, infarcts, and other abnormalities or signs of vascular injury. Data from subjects with abnormalities will be excluded from further analysis and they will be contacted and referred for a clinical scan. We expect less than 10% of scans to be excluded on this basis.

Cognitive Testing: Cognitive testing will be conducted on all subjects at baseline and at 12-week follow-up. The battery includes measures that we expect to be sensitive to subtle changes in cognitive function, as well as instruments that appear to have value in prospectively identifying individuals at risk for cognitive decline and/or dementia. Specifically, measures of working memory, memory recall, verbal fluency, executive function, and motor function will be used to detect early functional cognitive changes commonly seen in MCI.

The following battery of tests will take approximately 90 minutes (at both baseline and 12-week follow-up) to complete and will be administered during the afternoon to avoid diurnal effects: Auditory Consonant Trigrams; Benton Visual Retention Test 5th Edition, Boston Naming Test, Buschke-Fuld Selective Reminding Test, Delis Kaplan Executive Function System (DKEFS), Color-Word subtest, DKEFS Tower Test, DKEFS Trail Making Test, DKEFS Verbal Fluency subtest, Purdue Pegboard, Rey-Osterrieth Complex Figure Test, Taylor Complex Figure Task, Wechsler Abbreviated Scale of Intelligence, and the Wechsler Adult Intelligence Scale-3rd Edition.

Double-Blind Intervention: Following completion of the baseline assessments, volunteers will be randomly assigned to one of two 12- week interventions; double-blind placebo injection or liraglutide for 12 weeks. Subjects will be started on a subcutaneous morning dose of 0.6 mg, and this will be titrated to 1.2 mg after one week, and then titrated to 1.8 mg after one week and they will remain on this dose for the duration of the study (see Table 1). Subjects will be thoroughly instructed on how to self-administer the subcutaneous injection.

Any subject who cannot tolerate the highest dose, 1.8 mg due to side effects will be allowed to return to the 1.2 mg for the duration of the study. This dosing schedule is based on evidence that even the lowest dose has been shown to improve glycemic control in patients with type 2 diabetes, whereas the higher amounts have been used in studies in which estimates have been made of both insulin secretion and insulin sensitivity.

Subjects will have weekly phone visits with the clinical research coordinator during the first month, and then every two weeks for the remainder of the intervention. These calls will include an adverse events assessment. This assessment will be provided to the study's investigator and endocrinologist, Dr. Sun Kim, in order to determine patient dose. We will follow up on dose changes with patients within 48 hours to discuss these changes with them. Dr. Kim will meet with the patient if additional follow up on dosing is required.

After 12 weeks of treatment, all baseline evaluations will be repeated.

Anyone dropped from the study will not be replaced. All subjects will be unblinded upon completion of treatment or drop-out from the study. Open label treatment will not be offered.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be men and women between the ages of 50 and 70 yrs of age, with a BMI of 27 to 37 kg/m2 and at least 12 yrs of education.
* All subjects will be medically stable (i.e. no uncontrolled or poorly controlled medical illnesses), cognitively-intact as defined by Mini Mental Status Exam (MMSE) score of > 27, and will have adequate visual and auditory acuity to allow for cognitive testing.
* Metabolic function will be determined as impaired fasting glucose 100-125 mg/dL and/or impaired 2-hr glucose concentration 140-199 and <200mg/dL on 75-g oral glucose challenge.
* Also, half of all subjects will have a family history of dementia.

Exclusion Criteria:

* Diagnosis of possible or probable AD, MCI, or any other dementia; evidence of cognitive decline by MMSE score of <27 or self-reported significant decline in memory within the past year (per the Memory Function Questionnaire) (MFQ)
* History of Type I or Type II diabetes, or fasting plasma glucose > 126 mg/dL
* History of significant CVD or myocardial infarction; unstable cerebrovascular or pulmonary disease, gallstones, pancreatitis or cancer, multiple endocrine neoplasia (MEN) untreated hypothyroidism, unstable or untreated hypertension, anemia as determined by hematocrit < 30%
* Abnormal renal clearance as determined by the serum creatinine ³ 1.5 mg/d, hepatic dysfunction as determined by ALT > 2 times the upper limit of normal
* Presence of medications known to affect insulin action or insulin secretion
* Premature birth (which may affect MRI findings), history of neurological disorder (ischemic attacks, carotid bruits, or lacunes upon MRI scan), or evidence of neurologic or other physical illness that could produce cognitive deterioration; use of any drug that may significantly affect the OGTT results or cognitive testing results (specifically: cs)
* Drug or alcohol abuse or dependence within the past 6 months, positive urine toxicology screen for illicit substances at eligibility screening, history of mental illness, with the exception of past mood disorder, or evidence of acute depression as determined by a 17-item Hamilton Depression Rating Scale (HDRS-17) score of 8 or more.
* Participants with history of mood disorder must be in remission for at least 6 months prior to study entry.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Cognitive Outcomes | Change from Baseline to 3 months
  The following battery of tests will take approximately 90 minutes (at both baseline and 12-week follow-up) to complete and will be administered during the afternoon to avoid diurnal effects: Auditory Consonant Trigrams; Benton Visual Retention Test 5th Edition, Boston Naming Test, Buschke-Fuld Selective Reminding Test, Delis Kaplan Executive Function System (DKEFS), Color-Word subtest, DKEFS Tower Test, DKEFS Trail Making Test, DKEFS Verbal Fluency subtest, Purdue Pegboard, Rey-Osterrieth Complex Figure Test, Taylor Complex Figure Task, Wechsler Abbreviated Scale of Intelligence, and the Wechsler Adult Intelligence Scale-3rd Edition.
OGTT | Change from Baseline to 3 months
  Oral Glucose Tolerance Test (OGTT): After an overnight fast, subjects will be given a oral glucose challenge, wherein plasma glucose concentrations will be measured at baseline, T30min, T60min, T90min, and T120min after 75gm oral glucose load. Individuals with fasting glucose of 100-125 mg/dl and/or a 2-hour glucose of 140-199 mg/dL and less than 200 mg/dL will be eligible for study enrollment. OGTT will be repeated at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Rasgon, M.D., Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford Department of Psychiatry, Stanford, California, United States